CLINICAL TRIAL: NCT00835094
Title: A Randomized Trial Assessing the Chronobiology of Once Daily Administration of Mometasone Furoate DPI in Patients With Asthma
Brief Title: A Randomized Trial Assessing Once Daily Administration of Mometasone Furoate DPI in Asthmatics (Study P02177)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02177
Record Dates: First submitted 2008-10-30; First posted 2009-02-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morning (Experimental)
  Interventions: Device: Mometasone furoate
- Evening (Experimental)
  Interventions: Device: Mometasone furoate

INTERVENTIONS:
Device: Mometasone furoate — MF-DPI 400 mcg once daily in the morning for 12 weeks
  Other Names: Asmanex; SCH 32088
  Arms: Morning
Device: Mometasone furoate — MF-DPI 400 mcg once daily in the evening for 12 weeks
  Other Names: Asmanex; SCH 32088
  Arms: Evening

SUMMARY:
This will be an open-label, randomized, parallel-group comparison of mometasone furoate dry powder inhaler (MF-DPI) 400 mcg once daily administered in the morning vs. the evening for 12 weeks in subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (and their parent/guardian if the subject is <18) must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be >=12 years of age (unless restricted to an older age by local ethical committees or national health authorities), of either gender and any race.
* Subjects must have had a history of asthma for >=6 months.
* If the subject is taking inhaled corticosteroids, the daily dose must be <= the upper limit defined below:

  * budesonide <=800 mcg/day
  * triamcinolone acetonide <=800 mcg/day
  * beclomethasone dipropionate <=1000 mcg/day
  * fluticasone propionate <=500 mcg/day
  * flunisolide <=1000 mcg/day
* Women of childbearing potential must have a negative urine (hCG) pregnancy test on the day of randomization (Baseline visit).
* Women of childbearing potential (includes women who are <1 year postmenopausal) must be using an acceptable method of birth control (eg, hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (eg, hysterectomy or tubal ligation).
* Subjects must agree to inform their usual treating physician (if other than the study investigator) of their participation in this study.

Exclusion Criteria:

* Female subjects who are pregnant, breast-feeding, or are premenarcheal.
* Subjects who have required daily or alternate day oral corticosteroid treatment for more than a total of 14 days during the 6 months immediately prior to Visit 1, and/or subjects who have required a course of systemic corticosteroids within the previous month.
* Subjects who have had either an asthma exacerbation or a clinically relevant change in asthma medication within the last 4 weeks.
* Subjects who have been admitted to the hospital for asthma control within the previous 3 months or more than once within the previous 6 months.
* Subjects who have required ventilator support for respiratory failure secondary to their asthma within the last 5 years.
* Subjects who have used any investigational drug in the 30 days prior to Baseline, or subjects who have been treated with any investigational antibody for asthma in the 90 days prior to Baseline.
* Subjects who are allergic or have had an idiosyncratic reaction to corticosteroids.
* Subjects with any clinically significant disorder of the cardiovascular, neurologic, hematologic, gastrointestinal, cerebrovascular, or immunologic system, or respiratory disease other than asthma (eg, COPD), or any other disorder which may interfere with the study evaluations or affect subject safety.
* Subjects with a history of drug abuse, poor motivation, hypochondriasis, or any other emotional or intellectual problems that are likely to limit the validity of consent to participate in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2002-10-01 (Actual); Primary Completion 2003-07-01 (Actual); Study Completion 2003-07-01 (Actual)

PRIMARY OUTCOMES:
Between-treatment group comparisons (MF-DPI 400 mcg once daily in the morning compared to the evening) of daytime and nocturnal symptoms based on a 4 point scale. | 12 weeks
To compare the incidence of adverse events of MF-DPI 400 mcg once daily administered in the morning compared to the evening. | 12 weeks

SECONDARY OUTCOMES:
To assess morning vs. evening compliance with therapy. | 12 weeks
To assess subject satisfaction with the Twisthaler^TM device. | 12 weeks